CLINICAL TRIAL: NCT06791239
Title: Comparison of Thoracic Squeeze and Manual Diaphragmatic Release Technique on Respiratory Parameters and Functional Capacity in COPD Patients
Brief Title: Comparison of Thoracic Squeeze and Manual Diaphragmatic Release Technique in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Sabaoon Ijaz
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Thoracic squeeze technique; Manual diaphragmatic release technique; COPD; digital spirometry; functional capacity; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic squeeze technique (Experimental): The Thoracic Squeeze Technique is a manual physiotherapy intervention aimed at improving lung function, airway clearance, and respiratory mechanics. It involves the application of gentle, rhythmic compression to the chest wall during the exhalation phase of breathing, followed by a release. This technique can be performed with the patient in a sitting, semi-reclined, or supine position, depending on their condition and comfort level.
  Interventions: Other: Thoracic squeeze technique
- Manual Diaphragmatic release technique (Experimental): The Manual Diaphragmatic Release Technique is a soft tissue manipulation technique used to improve the mobility, function, and efficiency of the diaphragm. It is commonly applied in physiotherapy, particularly in respiratory, musculoskeletal, and manual therapy practices, to address breathing dysfunctions, postural imbalances, and associated pain or discomfort.
  Interventions: Other: Manual diaphragmatic release technique

INTERVENTIONS:
Other: Thoracic squeeze technique — The Thoracic Squeeze Technique is a manual therapy method used primarily in respiratory physiotherapy to improve lung expansion, enhance respiratory function, and facilitate secretion clearance in patients with respiratory conditions.
  Arms: Thoracic squeeze technique
Other: Manual diaphragmatic release technique — The Manual Diaphragmatic Release Technique is a soft tissue manipulation technique used to improve the mobility, function, and efficiency of the diaphragm. It is commonly applied in physiotherapy, particularly in respiratory, musculoskeletal, and manual therapy practices, to address breathing dysfunctions, postural imbalances, and associated pain or discomfort.
  Arms: Manual Diaphragmatic release technique

SUMMARY:
The goal of this randomized control trial is to evaluate and compare the efficacy of two physiotherapy techniques-Thoracic Squeeze Technique (TST) and Manual Diaphragmatic Release Technique (MDRT)-on improving respiratory parameters, functional capacity, and quality of life in patients with mild to moderate Chronic Obstructive Pulmonary Disease (COPD).

Objectives:

* Assess the impact of TST and MDRT on respiratory parameters (FEV1, FVC, FEV1/FVC ratio, and chest expansion).
* Compare the functional capacity outcomes of the two techniques using the 6-Minute Walk Test (6MWT).
* Evaluate the effects of TST and MDRT on patient wellbeing and daily life through the COPD Assessment Test (CAT).

Study Design:

The study involves 34 participants, divided into two groups (n=17 each) via sealed envelope randomization. Both groups will receive their respective interventions (TST or MDRT) alongside a standardized pulmonary rehabilitation protocol (pursed-lip breathing, diaphragmatic breathing, active cycle of breathing, and endurance exercises). The intervention will be conducted three times per week for three weeks.

Outcome Measures:

Primary outcomes include respiratory parameters assessed through spirometry and chest expansion using a measuring tape. Secondary outcomes include functional capacity (6MWT) and patient wellbeing (CAT scores). Baseline and post-intervention measures will be analyzed using SPSS, employing Mixed ANOVA to determine interaction effects.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic inflammatory condition of the respiratory system that progressively impairs airflow, leading to significant limitations in physical capacity and quality of life. COPD is a global health concern, being the third leading cause of death worldwide, with an increasing prevalence due to aging populations and environmental pollution. Despite advancements in pharmacological treatments, COPD management requires comprehensive rehabilitation strategies, particularly for improving respiratory function and functional capacity.

Two physiotherapy techniques, the Thoracic Squeeze Technique and Manual Diaphragmatic Release Technique, have been individually employed to address respiratory function in COPD patients. However, direct comparisons of their effectiveness on respiratory parameters, functional capacity, and overall quality of life are scarce. This study aims to evaluate and compare the effects of these techniques, combined with conventional pulmonary rehabilitation, to identify the more effective intervention for optimizing COPD treatment.

The trial will be conducted at Lady Reading Hospital, Peshawar, over six months following ethical approval.

This study will provide evidence-based insights into the relative efficacy of Thoracic Squeeze and Manual Diaphragmatic Release techniques. Findings will guide physiotherapists in optimizing rehabilitation protocols for COPD patients, improving respiratory function, functional capacity, and overall quality of life. Moreover, the research aims to contribute to the standardization of physiotherapy practices for COPD management, ensuring consistent and effective patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild or moderate COPD according to the GOLD criteria.GOLD 1: Mild FEV1 ≥ 80% predicted value, GOLD 2: Moderate FEV1 between 50% and 80% predicted value.
* Age between 40- 60 years.
* Both male and female.
* Patients who are willing to give voluntary consent to practice.

Exclusion Criteria:

* Patients with unstable hemodynamic parameters (arterial pressure <100mmHg Systolic and <60 mmHg diastolic blood pressure.
* Patients who have undergone recent 6 to 12 weeks cardio thoracic or abdominal surgery.
* Patients who have a recent history of chest wall or abdominal trauma; substantial chest wall deformity History of recent fractures and cognitive impairments.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Respiratory parameter FEV1/FVC ratio | 1 week
  The Gold standard tool used in the diagnosis of COPD is spirometry. In today GOLD guidelines the diagnosis of pulmonary function test based on a bronchodilator FEV1/FVC ratio of less than 0. 7.
Respiratory parameter Forced Expiratory Volume | 1 week
  Forced Expiratory Volume in 1 Second (FEV1 measures the volume of air that can be forcefully exhaled in the first second serving as an indicator of airway obstruction severity.
Respiratory parameter Forced Vital Capacity (FVC) | 1 week
  Forced Vital Capacity (FVC) the total volume of air exhale during a forced breath assessing overall lung capacity.
Functional capacity | 1 week
  Six Minute walk test:
  The 6-Minute Walk Test (6MWT) is a simple and practical test used to assess the functional exercise capacity of individuals. It measures the distance an individual can walk quickly on a flat hard surface in a period of six minutes. The test is commonly used in patients with chronic respiratory diseases such as COPD.

SECONDARY OUTCOMES:
Chest excursion | 1 week
  Chest excursion measurement is a simple clinical test used to assess the mobility of thoracic cage during respiration. This can be particularly useful in diagnosing and monitoring respiratory conditions such as COPD to measure lung expansion. Chest expansion will be measured at three levels; Upper Lobe: at the level of the fourth rib. Middle Lobe: at the level of the xiphoid process. Lower Lobe: at the level of the tenth rib.
Quality of life self-administered questionnaire | 3 weeks
  The COPD assessment test (CAT) is a self-administered questionnaire that consist of eight questions to explore different symptoms and impacts of COPD. .

CONTACTS AND LOCATIONS:
Overall Officials: Maria Naeem, DPT, MS-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Lady Reading Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braz Junior DS, Dornelas de Andrade A, Teixeira AS, Cavalcanti CA, Morais AB, Marinho PE. Whole-body vibration improves functional capacity and quality of life in patients with severe chronic obstructive pulmonary disease (COPD): a pilot study. Int J Chron Obstruct Pulmon Dis. 2015 Jan 12;10:125-32. doi: 10.2147/COPD.S73751. eCollection 2015. PMID 25624756